CLINICAL TRIAL: NCT00025545
Title: A Phase II Trial to Evaluate the Use of G-CSF-Mobilized Peripheral Blood Progenitor Cells as Hematopoietic Rescue in Patients With Acute Leukemia Undergoing Allografting From an Unrelated Donor
Brief Title: Filgrastim-Treated Donor Peripheral Stem Cell Transplantation in Treating Patients With Acute Leukemia</p>
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 1099.00; FHCRC-1099.00; NCI-H01-0078; CDR0000068972 (Registry Identifier: PDQ)
Record Dates: First submitted 2001-10-11; First posted 2003-06-20 (Estimated); Last update posted 2010-05-13 (Estimated); Status verified 2010-05

CONDITIONS: Leukemia
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; adult acute lymphoblastic leukemia in remission; childhood acute lymphoblastic leukemia in remission; acute undifferentiated leukemia; secondary acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute | interventions — Cyclophosphamide; Methotrexate; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Drug: cyclophosphamide
Drug: methotrexate
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Transplanted peripheral stem cells can sometimes be rejected by the body's tissues. Treating donor peripheral stem cells with filgrastim may increase the number of donor white blood cells. This may help to decrease the rejection of the transplanted cells in patients receiving them as treatment for acute leukemia.

PURPOSE: Phase II trial to study the effectiveness of filgrastim-treated donor peripheral stem cells in treating patients with acute leukemia who are undergoing peripheral stem cell transplantation.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether filgrastim (G-CSF)-mobilized allogeneic peripheral blood stem cell transplantation reduces the incidence of non-leukemic mortality in patients with acute leukemia.
* Determine the kinetics and durability of engraftment after treatment with this regimen in these patients.
* Determine the incidence and severity of acute and chronic graft-versus-host disease in patients treated with this regimen.
* Determine the leukemia-free survival of patients treated with this regimen.

OUTLINE: Donors receive filgrastim (G-CSF) subcutaneously (SC) on days -5 to -1. Donors then undergo leukapheresis on days -1 and 0.

Patients undergo total body irradiation twice daily on days -7 to -4. Patients receive 2 doses of intrathecal methotrexate per local guidelines between days -10 and -3. Patients also receive cyclophosphamide IV on days -3 and -2. Patients receive infusion of allogeneic peripheral blood stem cells on day 0.

PROJECTED ACCRUAL: A total of 5-60 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following diagnoses:

  * Primary acute leukemia beyond first remission
  * High-risk acute myelogenous leukemia
  * Acute lymphoblastic leukemia in first remission
* Must have HLA-matched donor identical for HLA-A, -B, and DRB1 alleles

  * No HLA-matched identical sibling or haploidentical relative incompatible for 0 or 1 HLA-A, -B, or -DRB1 loci on the non-shared haplotype
* No leukoencephalopathy

PATIENT CHARACTERISTICS:

Age:

* 55 and under

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* SGOT no greater than 2 times normal
* Hepatitis B surface antigen negative
* No prior hepatitis C

Renal:

* No impaired renal function
* Creatinine less than 2 times normal

Cardiovascular:

* No symptomatic cardiac disease

Pulmonary:

* No active pulmonary disease
* DLCO at least 60% predicted

Other:

* HIV negative
* No disease or other malignancy that severely limits life expectancy
* No severe or life-threatening infection within the past 2 weeks
* No history of septate fungal infection or disseminated candidiasis

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior bone marrow or peripheral blood stem cell transplantation

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy greater than 3,000 cGy to whole brain
* No prior radiotherapy of 1,500 cGy to chest or abdomen
* At least 6 months since prior involved-field radiotherapy to chest or abdomen

Surgery:

* Not specified

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1996-03; Primary Completion 2002-10 (Actual); Study Completion 2002-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Anasetti, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States